CLINICAL TRIAL: NCT03212976
Title: Assessment of the Clinical Efficacy of a Non-Invasive Measurement of Intracranial Pressure by Magnetic Resonance Phase Contrast Imaging
Brief Title: Clinical Efficacy of a Non-Invasive Measure of Intracranial Pressure
Acronym: MR-ICP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources are no longer available
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ronald Benveniste, Associate Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20170130
Record Dates: First submitted 2017-06-29; First posted 2017-07-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Intracranial Pathology; Intracranial Hypertension
Keywords: Non-Invasive; Magnetic Resonance Imaging; Ventricular catheters
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Phase 1 (Other): Patients with an intracranial pressure monitor will undergo phase contrast magnetic resonance imaging to measure their ICP.
  Interventions: Procedure: Phase contrast magnetic resonance imaging
- Study Phase 2 (Other): Patients with shunts or CSF access devices such as Ommaya reservoir, etc will undergo phase contrast magnetic resonance imaging
  Interventions: Procedure: Phase contrast magnetic resonance imaging

INTERVENTIONS:
Procedure: Phase contrast magnetic resonance imaging — Phase-contrast magnetic resonance imaging will be done to assess intracranial pressure

SUMMARY:
This study is designed to evaluate the accuracy of a non-invasive method phase-contrast magnetic resonance imaging (MR-ICP) for assessing intracranial pressure (Phase 1).

To perform second phase contrast imaging to evaluate the patency and flow of ventricular catheters after MR-ICP imaging (Phase 2).

DETAILED DESCRIPTION:
The study will be divided into 2 phases. In Phase 1, patients with an intracranial pressure monitor will be recruited to the study, while in Phase 2, patients with shunts or Cerebral Spinal Fluid (CSF) access devices (Ommaya, reservoir, etc.) will be eligible for the study.

Two separate groups of patients will be recruited to each phase of the study. Each phase of the study will involve MR-ICPs. The MR-ICP is an extra 5-10 minute sequence at the end of a MRI that assesses the pressure in the head. The MRI will take scans of the brain during different phases of the cardiac cycle and will assess the volume changes while the patient is lying flat. The pressure in the head will be estimated based on these calculations. This estimate will be compared to the pressure in the head as determined by the ICP monitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for a MRI by Attendings in the Department of Neurological Surgery at the University of Miam with intracranial pathology with external ventricular drains (EVDs) or intracranial bolts placed for hydrocephalus or intracranial hypertension. Bolts must be placed prior to enrollment in the study to avoid any alterations in standard procedure
* All pathological entities that produce intracranial hypertension will be included (trauma, tumor, vascular, infectious, inflammatory, etc).
* Patients must undergo a MRI for another clinically indicated reason (diagnosis, surveillance, cervical MRI clearance, prognosis, etc).
* English and Spanish-speaking patients

Exclusion Criteria:

* Unable to obtain MRI due to prior implants, metallic material, inability to sit still
* Refractory intracranial hypertension (not controlled with medications, surgery, or EVD)
* Unable to obtain informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Intracranial Pressure Measurement | 1 day
  Ratio of intracranial volume
Patency of ventricular catheters | 7 days
  Patency of ventricular catheters will be measured using multi-voxel MRI-ICP to qualitatively assess presence of CSF flow.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Benveniste, MD, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: No